CLINICAL TRIAL: NCT00955968
Title: IMPAACT 1077HS: HAART Standard Version of the Promoting Maternal and Infant Survival Everywhere (PROMISE) Study
Brief Title: IMPAACT 1077HS: Examining Benefits of HAART Continuation in Postpartum Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 1077HS; U01AI068632 (NIH)
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: HIV Infection
Keywords: HIV Infection; HAART; Maternal Health
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continue HAART (Experimental): Continue receiving HAART within 0-42 days after delivery or other pregnancy outcome.
  Interventions: Drug: Highly active antiretroviral therapy (HAART)
- Stop HAART (Active Comparator): Stop receiving HAART within 0-42 days after delivery or other pregnancy outcome and resume HAART when protocol specified criteria were met.
  Interventions: Drug: Highly active antiretroviral therapy (HAART)

INTERVENTIONS:
Drug: Highly active antiretroviral therapy (HAART) — A combination of three or more HIV medications belonging to two or more drug classes.
  The preferred study-supplied HAART regimen was lopinavir/ritonavir (LPV/RTV) plus fixed dose combination tenofovir/emtricitabine (TDF/FTC). Additional ARVs provided for use in this study included fixed dose combination lamivudine/zidovudine (3TC/ZDV), lamivudine (3TC), zidovudine (ZDV), tenofovir (TDF), fixed dose combination tenofovir/emtricitabine/rilpivirine (TDF/FTC/RPV), didanosine (ddI), atazanavir (ATV), raltegravir (RAL), and ritonavir (RTV). While LPV/RTV plus TDF/FTC was the preferred study-supplied regimen, the study clinicians in conjunction with participants would determine the optimal drug combination for each participant.

SUMMARY:
This study was a randomized strategy trial conducted among women who received highly active antiretroviral therapy (HAART) during pregnancy for purposes of prevention of mother-to-child transmission (PMTCT) of HIV but did not otherwise meet criteria to initiate HAART for their own health. The study was designed to determine whether continuation of HAART after delivery or other pregnancy outcome reduced morbidity and mortality compared to discontinuation and re-initiation of HAART when protocol specified criteria were met.

DETAILED DESCRIPTION:
This randomized strategy trial addressed therapeutic questions for women from regions where antepartum HAART for PMTCT (for all CD4+ cell counts) and postpartum formula feeding is standard of care, and who also had both a pre-HAART CD4+ cell count >400 cells/mm^3 and a screening (on-HAART) CD4+ cell count > 400 cells/mm^3. For these women, the objectives related to the relative efficacy and safety of continuing HAART (when it is no longer used for PMTCT) versus discontinuing HAART.

Potential participants were identified/recruited and consented during pregnancy or after delivery or other pregnancy outcome. Study-specific screening was initiated in the third trimester or after pregnancy outcome. Women who were screened for the study were counseled to continue their HAART until they were randomized.

Randomization would occur within 0-42 days after pregnancy outcome. Women who did not carry their pregnancy to the third trimester but otherwise meet study eligibility criteria could be enrolled.

Participants were randomized to one of the two study arms:

Arm A: Continuation of HAART Arm B: Discontinuation of HAART and resume HAART when protocol-specified criteria were met

Participants were to be followed until 84 weeks after the last participant was randomized.

Key evaluations were conducted at Screening, Entry, post entry visits were scheduled to take place 4 weeks after entry, 12 weeks after entry, and every 12 weeks thereafter. Key evaluations included physical examinations, clinical assessments, and blood collection.

On 7 July 2015, the study sites received formal communications regarding the results of the Strategic Timing of Antiretroviral Treatment (START) study and associated changes were implemented to the 1077HS study in response to these results. All sites were instructed that all women in the 1077HS study were to be informed of the START study results and that antiretroviral therapy (ART) was recommended for all women based on the START study results.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18 years or who had attained the minimum age of independent consent, as defined by the local Institutional Review Board (IRB), and were willing and able to provide written informed consent Additionally, at sites with IRB approval to enroll younger participants, women age 16-17 years who were willing and able to provide written assent and whose parent or legal guardian was willing and able to provide written informed consent
* Confirmed HIV infection, documented by positive results from two samples collected at different time points prior to study entry, using protocol-specified tests (see protocol for more details)
* Documentation of hepatitis B surface antibody (HBsAb) status and hepatitis B surface antigen (HBsAg) status (if antibody was negative) within 12 months prior to study entry
* Within 0-42 days after pregnancy outcome
* Antiretroviral treatment naïve, defined as < 14 days of one or more antiretroviral agents, prior to therapy initiated during current pregnancy
* Receipt of at least four weeks of HAART prior to study entry, at least two weeks of which must have been prior to pregnancy outcome (up to seven consecutive days of missed therapy is permitted)
* CD4+ cell count ≥ 400 cells/mm^3 on a specimen obtained within 120 days prior to initiation of HAART for current pregnancy
* CD4+ cell count ≥ 400 cells/mm^3 on a specimen obtained on HAART and within 45 days prior to study entry
* The following laboratory values on a specimen obtained within 45 days prior to study entry:

  * Absolute neutrophil count ≥ 750/mm^3
  * Hemoglobin ≥ 7.0 g/dL
  * Platelet count ≥ 50,000/mm^3
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 2.5 x ULN
* Estimated creatinine clearance of ≥ 60mL/min within 45 days prior to entry using the Cockcroft-Gault formula
* Intent to remain in current geographical area of residence for the duration of the study
* Willingness to attend study visits as required by the study

Exclusion Criteria:

* Previous participation in PROMISE (P1077BF - NCT01061151)
* Clinical indication for HAART including any World Health Organization (WHO) Clinical Stage 3 or 4 condition, prior or current tuberculosis disease (a positive (Purified protein Derivative) PPD test alone was not considered exclusionary), and/or any other clinical indication per country-specific treatment guidelines
* Clinically significant illness or condition requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Social or other circumstances which, in the opinion of the site investigator, would hinder long-term follow up
* Use of any prohibited medications within 14 days prior to study entry (refer to the study MOP for a list of prohibited medications)
* Current compulsory detention (involuntary incarceration) in a correctional facility, prison, or jail for legal reasons or compulsory detention in a medical facility for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Currently breastfeeding or planning to breastfeed
* Current documented conduction heart defect (specialized assessments to rule out this condition were not required; a heart murmur alone and/or type 1 second-degree atrioventricular block (also known as Mobitz I or Wenckebach) was not considered exclusionary)
* Known evidence of HBV DNA levels >2000 IU/mL (approximately 10,000 copies/mL) in the presence of elevated (grade 1 and higher) ALT (HBV DNA testing was not required for study screening or enrollment but was considered to determine whether treatment for HBV was indicated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Currier, MD, MS, Study Chair — University of California, Los Angeles
Locations (50):
- United States (26):
  - University of Southern California MCA Center (5048), Alhambra, California
  - David Geffen School of Medicine at UCLA (5112), Los Angeles, California
  - UCSD Mother-Child-Adolescent HIV Program (4601), San Diego, California
  - Harbor (UCLA) Medical Center (5045), Torrance, California
  - University of Colorado (5052), Aurora, Colorado
  - Howard University (5044), Washington D.C., District of Columbia
  - Georgetown University (1008), Washington D.C., District of Columbia
  - Washington Hospital Center (5023), Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center (5055), Fort Lauderdale, Florida
  - University of Florida at Jacksonville (5051), Jacksonville, Florida
  - University of Miami Pediatric/Perinatal Clinical Research Site (4201), Miami, Florida
  - University of South Florida at Tampa (5018), Tampa, Florida
  - Ann & Robert H Lurie Children's Hospital of Chicago (4001), Chicago, Illinois
  - Tulane University (5095), New Orleans, Louisiana
  - Johns Hopkins University School of Medicine (5092), Baltimore, Maryland
  - Boston Medical Center (5011), Boston, Massachusetts
  - Wayne State University/Children's Hospital of Michigan (5041), Detroit, Michigan
  - Metropolitan Hospital (5003), New York, New York
  - SUNY Stony Brook University Medical Center (5040), Stony Brook, New York
  - Bronx-Lebanon Hospital Center (5114), The Bronx, New York
  - Jacobi Medical Center (5013), The Bronx, New York
  - Duke University Medical Center (4701), Durham, North Carolina
  - Pitt CRS (1001), Pittsburgh, Pennsylvania
  - St Jude Children's Research Hospital (6501), Memphis, Tennessee
  - Baylor College of Medicine Texas Children's Hospital (3801), Houston, Texas
  - Seattle Children's Hospital (5017), Seattle, Washington
- Hospital General de Agudos (5082), Buenos Aires, Argentina
- Botswana (2):
  - Gaborone Prevention/Treatment Clinical Research Site (12701), Gaborone
  - Molepolole Prevention/Treatment Clinical Research Site (12702), Gaborone
- Brazil (8):
  - School of Medicine, University of Minas Gerais - FUNDEP (5073), Belo Horizonte
  - University Caxias do Sul (5084), Caxias do Sul
  - Hospital Nossa Senhora da Conceicao (5117), Porto Alegre
  - Hospital Santa Casa (5098), Porto Alegre
  - Hospital dos Servidores do Estado (5072), Rio de Janeiro
  - Hospital Geral De Nova Igaucu (5097), Rio de Janeiro
  - Instituto de Puericultura E Pediatria Martagao Geseira - FUJB (5071), Rio de Janeiro
  - Ribeirao Preto Medical School, University of Sao Paulo (5074), São Paulo
- Guangxi Center for HIV/AIDS Prevention and Control (30274), Nanning, Guangxi, China
- Les Centres GHESKIO (30022), Port-au-Prince, Haiti
- Peru (2):
  - IMPACTA Barranco Clinical Research Site (11301), Lima
  - IMPACTA San Miguel Clinical Research Site (11302), Lima
- Puerto Rico (2):
  - San Juan City Hospital (5031), San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research Program (6601), San Juan
- Thailand (7):
  - Siriraj Hospital Mahidol University CRS (5115), Bangkok, Ratchathewi,
  - Bhumibol Adulyadej Hospital (5124), Bangkok
  - Prapokklao Hospital (5123), Chanthaburi
  - Chiang Mai University (31784), Chiang Mai
  - Chiang Rai Regional Hospital (5116), Chiang Rai
  - Chonburi Hospital (5125), Chon Buri
  - Phayao Provincial Hospital (5122), Phayao

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 with Clarification dated August 2009, which can be found on the DAIDS RSC Web site: http://rsc.tech-res.com
- [Background] Manual for Expedited Reporting of Adverse Events to DAIDS, Version 2.0, January 2010.
- [Derived] Currier JS, Britto P, Hoffman RM, Brummel S, Masheto G, Joao E, Santos B, Aurpibul L, Losso M, Pierre MF, Weinberg A, Gnanashanmugam D, Chakhtoura N, Klingman K, Browning R, Coletti A, Mofenson L, Shapiro D, Pilotto J; 1077HS PROMISE Team. Randomized trial of stopping or continuing ART among postpartum women with pre-ART CD4 >/= 400 cells/mm3. PLoS One. 2017 May 10;12(5):e0176009. doi: 10.1371/journal.pone.0176009. eCollection 2017. PMID 28489856
- See also: Related Info — http://www.impaactnetwork.org/studies/1077HS.asp
- See also: WHO Case Definitions of HIV for Surveillance and Revised Clinical Staging and Immunological Classification of HIV-related Disease in Adults and Children (World Health Organization 2007). — http://apps.who.int/iris/handle/10665/43699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 1653 participants randomized to the study with enrollments from the US, Argentina, Botswana, Brazil, China, Haiti, and Thailand. The first participant was randomized on January 2010. The last participant was randomized in November 2014.
Pre-assignment Details: There were 1917 participants screened for the study, 264 of these failed screening and were not enrolled. The most common reasons for screening failure were CD4 cell count out of range, did not return for consent, test results unavailable on protocol specified time frame, not willing to participate, and not willing to remain on antiretrovirals.
Period: Overall Study
Arm/Group | Continue HAART | Stop HAART
Started | 828 | 825
Completed | 691 | 699
Not Completed | 137 | 126
Not completed — Death | 2 | 4
Not completed — Withdrawal by Subject | 35 | 31
Not completed — Lost to Follow-up | 45 | 39
Not completed — Site closed | 55 | 52

BASELINE CHARACTERISTICS:
Population: All the participants who were randomized to the study with the exception of one participant who was excluded as she withdrew from the study on the day she was randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Continue HAART | Stop HAART | Total
Number analyzed (Participants) | 827 | 825 | 1652
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 18 | 36
  Between 18 and 65 years | 809 | 807 | 1616
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [23 to 32] | 28 [24 to 32] | 28 [23 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 827 | 825 | 1652
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 32 | 29 | 61
  Argentina | 20 | 25 | 45
  United States | 72 | 77 | 149
  Botswana | 230 | 227 | 457
  China | 52 | 52 | 104
  Brazil | 259 | 255 | 514
  Thailand | 156 | 151 | 307
  Peru | 6 | 9 | 15
Race/Ethnicity [Count of Participants; unit: Participants]
  Asian | 209 | 203 | 412
  Black or African American | 58 | 58 | 116
  White | 123 | 127 | 250
  American Indian | 1 | 1 | 2
  Alaskan Native | 0 | 1 | 1
  Black African | 230 | 227 | 457
  Black of African origin | 77 | 70 | 147
  Mestizo | 6 | 8 | 14
  Mixed Black | 73 | 76 | 149
  Mixed native | 0 | 4 | 4
  Native (native Brazilian-Xavante/Kaigang/Guarani) | 1 | 1 | 2
  Other | 31 | 31 | 62
  Subject does not know | 4 | 2 | 6
  Race not available to clinic | 14 | 16 | 30
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] — Population: Baseline weight and height measure were not completed for some participants
  kg/m^2
    number analyzed (Participants) | 812 | 801 | 1613
    (all) | 24.4 [21.7 to 28.0] | 24.6 [21.8 to 28.3] | 24.5 [21.8 to 28.1]
WHO stage at entry [Count of Participants; unit: Participants] — Clinical staging of HIV/AIDS by WHO definitions (WHO, 2007). Staging is based on clinical findings that guide the diagnosis, evaluation, and management of HIV/AIDS. Clinical stages are categorized as 1 through 4, progressing from primary HIV infection to advanced HIV/AIDS. These stages are defined by specific clinical conditions or symptoms as described in the reference (see the References in the Protocol Section). Population: Baseline WHO staging criteria was not completed for some participants.
  Participants
    number analyzed (Participants) | 827 | 823 | 1650
    Clinical Stage I | 810 | 811 | 1621
    Clinical Stage II | 16 | 11 | 27
    Clinical Stage III | 1 | 1 | 2
Duration of Antiretroviral therapy (ART) prior to study entry [Median (Inter-Quartile Range); unit: weeks] | 17 [11 to 23] | 17 [11 to 23] | 17 [11 to 23]
ART regimen prior to entry [Count of Participants; unit: Participants] — PI - Protease Inhibitor, NNRTI - Non Nucleoside Reverse Transcriptase Inhibitor, EFV - Efavirenz, NVP - Nevirapine, RPV - Rilpivirine, NRTI - Nucleoside Reverse Transcriptase Inhibitor, II - Integrase Inhibitor
  Participants
    HAART including boosted PI | 629 | 612 | 1241
    HAART including non-boosted PI | 12 | 16 | 28
    HAART including NNRTI [EFV] | 180 | 172 | 352
    HAART including NNRTI [NVP] | 4 | 8 | 12
    HAART including NNRTI [RPV] | 1 | 1 | 2
    HAART including NNRTI and PI | 1 | 0 | 1
    Three or more NRTIs | 3 | 11 | 14
    Zero NRTIs | 0 | 1 | 1
    HAART including II | 4 | 4 | 8
    HAART including PI and II | 2 | 0 | 2
Hepatitis B surface antigen [Count of Participants; unit: Participants] — Population: Baseline Hepatitis B surface antigen was not obtained for some participants
  Participants
    Positive: number analyzed (Participants) | 821 | 819 | 1640
    Positive | 29 | 28 | 57
    Negative: number analyzed (Participants) | 821 | 819 | 1640
    Negative | 771 | 768 | 1539
    Indeterminate: number analyzed (Participants) | 821 | 819 | 1640
    Indeterminate | 1 | 0 | 1
    Not obtained, Hep B antibody +ve: number analyzed (Participants) | 821 | 819 | 1640
    Not obtained, Hep B antibody +ve | 20 | 23 | 43
Hepatitis B surface antibody [Count of Participants; unit: Participants] — Population: Baseline Hepatitis B surface antibody was not obtained for some participants
  Participants
    Positive: number analyzed (Participants) | 826 | 823 | 1649
    Positive | 263 | 248 | 511
    Negative: number analyzed (Participants) | 826 | 823 | 1649
    Negative | 424 | 425 | 849
    Indeterminate: number analyzed (Participants) | 826 | 823 | 1649
    Indeterminate | 1 | 2 | 3
    Not obtained, Hep B antibody +ve: number analyzed (Participants) | 826 | 823 | 1649
    Not obtained, Hep B antibody +ve | 138 | 148 | 286
CD4+ cell count on ART [Median (Inter-Quartile Range); unit: cells/mm^3] — CD4+ cell count was evaluated at screening
  cells/mm^3 | 696 [575 to 870] | 695 [575 to 868] | 696 [575 to 869]
Pre-ART CD4+ cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 550 [461 to 682] | 548 [463 to 677] | 549 [462 to 680]
Plasma HIV Viral Load [Count of Participants; unit: Participants] — Population: Baseline Plasma HIV viral load was not obtained for some participants
  Participants
    < 400 copies/ml: number analyzed (Participants) | 822 | 819 | 1641
    < 400 copies/ml | 744 | 742 | 1486
    400 - <1000 copies/ml: number analyzed (Participants) | 822 | 819 | 1641
    400 - <1000 copies/ml | 30 | 24 | 54
    1000- <10000 copies/ml: number analyzed (Participants) | 822 | 819 | 1641
    1000- <10000 copies/ml | 32 | 29 | 61
    10000-<100000 copies/ml: number analyzed (Participants) | 822 | 819 | 1641
    10000-<100000 copies/ml | 15 | 24 | 39
    >=100000 copies/ml: number analyzed (Participants) | 822 | 819 | 1641
    >=100000 copies/ml | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of AIDS - Defining Illness, Serious Non-AIDS Defining, Cardiovascular, Renal, Hepatic Event, or Death
Description: AIDS defining illness, serious non-AIDS defining cardiovascular, renal, or hepatic event, or death refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: From study entry to study termination, all participants were followed until July 7, 2015 (an average of 125 weeks of follow-up).
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 0.21 [0.16 to 0.27] | 0.31 [0.25 to 0.38]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.54, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.19 to 2.40] — HR reflects Continue HAART : Stop HAART

2. Secondary Outcome: Incidence Rate of AIDS - Defining Illness
Description: AIDS defining illness, refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 0.10 [0.08 to 0.14] | 0.15 [0.12 to 0.19]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.66, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.11 to 4.01] — HR reflects Continue HAART : Stop HAART

3. Secondary Outcome: Incidence Rates of Serious Non- AIDS Defining Cardiovascular, Renal or Hepatic Event
Description: Serious non - AIDS defining cardiovascular, renal, or hepatic event, or death refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Incidence Rate of Deaths
Description: The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 0.10 [0.08 to 0.14] | 0.20 [0.17 to 0.25]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.44, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.09 to 2.81] — HR reflects Continue HAART : Stop HAART

5. Secondary Outcome: Incidence Rate of HIV/AIDS Related Events
Description: HIV/AIDS related events refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 1.32 [1.07 to 1.62] | 1.42 [1.16 to 1.73]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.79, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.54 to 1.60] — HR reflects Continue HAART : Stop HAART

6. Secondary Outcome: Incidence Rate of HIV/AIDS Related Events or Death
Description: HIV/AIDS related events or death refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 1.42 [1.16 to 1.75] | 1.57 [1.30 to 1.91]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.71, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.54 to 1.52] — HR reflects Continue HAART : Stop HAART

7. Secondary Outcome: Incidence Rate of HIV/AIDS Related Events or WHO Clinical Stage 2 or 3 Events
Description: HIV/AIDS related events or WHO Clinical Stage 2 or 3 events refers to illness/diagnoses listed in Appendix II of the protocol. These events were reviewed and confirmed by an Endpoint review group. The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 3.09 [2.52 to 3.79] | 5.37 [4.60 to 6.28]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p < 0.001, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.42 to 0.80] — HR reflects Continue HAART : Stop HAART

8. Secondary Outcome: Incidence Rate of Grade 2 and Above Toxicity
Description: The toxicity events included all grade 2 and higher hematology or chemistry events and grade 3 or 4 sign or symptoms. These events were graded using the Division of AIDS (DAIDS AE Grading Table), Version 1.0, December 2004, Clarification August 2009, which is available on the RSC website (http://rsc.tech-res.com). The incidence rate was obtained by using the Kaplan-Meier method.
Time Frame: All laboratory measures were done at entry,4 and 12 weeks after, and then every 3 months until study end. Signs and Symptoms were recorded from study entry to study end. All were followed until July 7, 2015 (an average of 125 weeks of follow-up)
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Number (95% Confidence Interval); unit: New cases per 100 person - years
Groups:
- Continue HAART: Participants would continue receiving HAART after delivery or other pregnancy outcome.
  Highly active antiretroviral therapy (HAART): A combination of three or more HIV medications belonging to two or more drug classes
- Stop HAART: Participants would stop receiving HAART after delivery or other pregnancy outcome and resume HAART when protocol-specified criteria were met.
  Highly active antiretroviral therapy (HAART): A combination of three or more HIV medications belonging to two or more drug classes
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
New cases per 100 person - years | 18.4 [15.7 to 21.4] | 15.6 [13.2 to 18.4]
Statistical Analysis 1: Comparison: Continue HAART vs Stop HAART; Test type: Superiority; p = 0.10, Log Rank — 5% alpha level and 2-sided test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.03]

9. Secondary Outcome: Incidence Rate of Cardiovascular or Other Metabolic Events
Description: This outcome was intended as an exploratory analyses and was not included in the primary analyses conditional on primary results and funding. Given the results of the primary analyses it was decided that this outcome was no longer scientifically important. No resources and funding was allocated by NIH.
Time Frame: as for outcome 1
Population: This outcome was intended as an exploratory analyses and was not included in the primary analyses conditional on primary results and funding. Given the results of the primary analyses it was decided that this outcome was no longer scientifically important. No resources and funding was allocated by NIH.
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Incidence Rate of Other Targeted Medical Conditions
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 9
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence Rate of Any Condition Outlined in Appendix II of Protocol or Death
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 9
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Virologic Failure (VF) Participants With HIV Resistance in the Continue HAART Arm
Description: VF was defined as two successive measurements of HIV-1 RNA above 1000 copies/ml at or after 24 weeks of HAART. HIV drug resistance was defined using the Stanford database (Version 6.2)
Time Frame: At time of confirmation of VF. HIV-1 RNA testing to identify VF was done at week 4, 12, 24, and every 12 weeks thereafter until study end at an average of 125 weeks. If HIV-1 RNA was above 1000 copies/ml, confirmatory testing was done within 4 weeks.
Population: 156 women who were VFs had antiretroviral drug resistance testing performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART
Number analyzed (Participants) | 156
Participants | 19

13. Secondary Outcome: Medication Adherence - Last Time Missed Medications
Description: Medication adherence was evaluated by a self reported questionnaire. The number of participants who indicated predefined choice is provided.
Time Frame: week 0, 48 and 96
Population: Participants in the Continue HAART arm who had evaluations done at the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART
Number analyzed (Participants) | 672
Participants
  Week 0: Never skipped medications | 489
  Week 0: More than 1 month ago | 60
  Week 0: Within the past 4 weeks | 123
  Week 48: number analyzed (Participants) | 652
  Week 48: Never skipped medications | 411
  Week 48: More than 1 month ago | 97
  Week 48: Within the past 4 weeks | 144
  Week 96: number analyzed (Participants) | 638
  Week 96: Never skipped medications | 399
  Week 96: More than 1 month ago | 92
  Week 96: Within the past 4 weeks | 147

14. Secondary Outcome: Medication Adherence - How Closely Followed Schedule
Description: as for outcome 13
Time Frame: week 0, 48 and 96
Population: Participants in the Continue HAART arm who had evaluations done at the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART
Number analyzed (Participants) | 673
Participants
  Week 0: Never | 23
  Week 0: Some of the time | 130
  Week 0: All of the time | 520
  Week 48: number analyzed (Participants) | 651
  Week 48: Never | 17
  Week 48: Some of the time | 173
  Week 48: All of the time | 461
  Week 96: number analyzed (Participants) | 637
  Week 96: Never | 25
  Week 96: Some of the time | 153
  Week 96: All of the time | 459

15. Secondary Outcome: Medication Adherence - How Often Follow Instructions
Description: as for outcome 13
Time Frame: week 0, 48 and 96
Population: Participants in the Continue HAART arm who had evaluations done at the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART
Number analyzed (Participants) | 667
Participants
  Week 0: Never | 10
  Week 0: Some of the time | 52
  Week 0: All of the time | 166
  Week 0: No special instructions | 439
  Week 48: number analyzed (Participants) | 650
  Week 48: Never | 6
  Week 48: Some of the time | 61
  Week 48: All of the time | 194
  Week 48: No special instructions | 389
  Week 96: number analyzed (Participants) | 637
  Week 96: Never | 8
  Week 96: Some of the time | 74
  Week 96: All of the time | 190
  Week 96: No special instructions | 365

16. Secondary Outcome: Medication Adherence - Missed Dose Within Past 4 Days
Description: as for outcome 13
Time Frame: week 0, 48 and 96
Population: Participants in the Continue HAART arm who had evaluations done at the respective weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART
Number analyzed (Participants) | 653
Participants
  Week 0: No | 592
  Week 0: Yes | 61
  Week 48: number analyzed (Participants) | 635
  Week 48: No | 564
  Week 48: Yes | 71
  Week 96: number analyzed (Participants) | 621
  Week 96: No | 544
  Week 96: Yes | 77

17. Secondary Outcome: Quality of Life - General Health Outcome
Description: Quality of Life was evaluated by a self reported questionnaire. The number of participants who indicated predefined choice is provided.
Time Frame: week 0, 48 and 96
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
Participants
  week 0: number analyzed (Participants) | 823 | 818
  week 0: Excellent | 160 | 164
  week 0: Very good | 262 | 269
  week 0: Good | 327 | 333
  week 0: Fair | 71 | 51
  week 0: Poor | 3 | 1
  week 48: number analyzed (Participants) | 701 | 701
  week 48: Excellent | 172 | 185
  week 48: Very good | 250 | 229
  week 48: Good | 222 | 238
  week 48: Fair | 52 | 48
  week 48: Poor | 5 | 1
  week 96: number analyzed (Participants) | 500 | 504
  week 96: Excellent | 131 | 134
  week 96: Very good | 179 | 178
  week 96: Good | 165 | 157
  week 96: Fair | 23 | 34
  week 96: Poor | 2 | 1

18. Secondary Outcome: Quality of Life (QoL) - Health Rating Score
Description: QoL - health rating score was evaluated by a self reported questionnaire. Health rating score of 0 was indicative of death or worst possible health and a score of 100 was being in perfect or best possible health and the mean of score is calculated. Higher scores indicate better Quality of Life (QoL). The range is 0-100 units on a scale
Time Frame: week 0, 48 and 96
Population: All participants except one who was excluded as she withdrew from study on the day she was randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 827 | 825
units on a scale
  week 0: number analyzed (Participants) | 819 | 820
  week 0 | 82.7 (15.7) | 83.0 (15.1)
  week 48: number analyzed (Participants) | 703 | 702
  week 48 | 85.3 (14.7) | 85.4 (14.0)
  week 96: number analyzed (Participants) | 501 | 504
  week 96 | 86.2 (14.1) | 86.3 (14.0)

19. Secondary Outcome: Changes in Plasma Concentrations of Inflammatory and Thrombogenic Markers
Description: This outcome was intended as an exploratory analyses and was not included in the primary analyses conditional on primary results and funding. This outcome required additional funding for laboratory testing which was not available and so this outcome is not reported.
Time Frame: Measured at baseline, after 4 and 12 weeks, and then every 6 months until study termination. All participants were followed until July 7, 2015 (an average of 125 weeks of follow-up).
Population: This outcome was intended as an exploratory analyses and was not included in the primary analyses conditional on primary results and funding. This outcome required additional funding for laboratory testing which was not available and so this outcome is not reported.
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Cost Effectiveness and Feasibility of Treatment Models
Description: This outcome was intended as an exploratory analyses and was not included in the primary analyses. Given the results of the primary analyses and changes in WHO guidelines to recommend lifelong antiretroviral therapy, the protocol team decided that this outcome was no longer scientifically important. No resources and funding was allocated by NIH.
Time Frame: Measured at baseline, after 4 - 12 and 24 weeks, and then every 6 months until study termination. All participants were followed until July 7, 2015 (an average of 125 weeks of follow-up).
Population: This outcome was intended as an exploratory analyses and was not included in the primary analyses. Given the results of the primary analyses and changes in WHO guidelines to recommend lifelong antiretroviral therapy, the protocol team decided that this outcome was no longer scientifically important. No resources and funding was allocated by NIH.
Arm/Group | Continue HAART | Stop HAART
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From study entry to off study date (an average of 125 weeks of follow-up).
Description: The study protocol required reporting of all new diagnoses, signs/symptoms and laboratory events of >=Grade 3 (with exceptions to all grades of creatinine and all grade >=2 renal, hematologic, and hepatic abnormalities), and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used.
Groups:
- Stop HAART: Participants would stop receiving HAART after delivery or other pregnancy outcome and resume when protocol-specified criteria were met.
  Highly active antiretroviral therapy (HAART): A combination of three or more HIV medications belonging to two or more drug classes
Arm/Group | Continue HAART | Stop HAART
All-Cause Mortality (participants affected / at risk) | 2/827 | 4/825
Serious Adverse Events (participants affected / at risk) | 10/827 | 3/825
Other Adverse Events (participants affected / at risk) | 778/827 | 765/825
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continue HAART (N=827) | Stop HAART (N=825)
Endophthalmitis (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Ergot poisoning (Injury, poisoning and procedural complications) | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continue HAART (N=827) | Stop HAART (N=825)
Diarrhoea (Gastrointestinal disorders) | 65 | 38
Nausea (Gastrointestinal disorders) | 54 | 48
Vomiting (Gastrointestinal disorders) | 46 | 37
Acute sinusitis (Infections and infestations) | 31 | 60
Bacterial vaginosis (Infections and infestations) | 62 | 67
Cervicitis (Infections and infestations) | 62 | 48
Tonsillitis (Infections and infestations) | 50 | 71
Urinary tract infection (Infections and infestations) | 37 | 48
Viral upper respiratory tract infection (Infections and infestations) | 60 | 53
Vulvovaginal candidiasis (Infections and infestations) | 58 | 97
Alanine aminotransferase increased (Investigations) | 70 | 71
Aspartate aminotransferase increased (Investigations) | 51 | 44
Blood bicarbonate decreased (Investigations) | 49 | 61
Blood bilirubin increased (Investigations) | 148 | 57
Blood cholesterol increased (Investigations) | 527 | 500
Blood glucose abnormal (Investigations) | 58 | 51
Blood glucose decreased (Investigations) | 121 | 91
Blood glucose increased (Investigations) | 117 | 123
Blood phosphorus decreased (Investigations) | 103 | 76
Blood sodium decreased (Investigations) | 88 | 100
Haemoglobin decreased (Investigations) | 68 | 63
Low density lipoprotein increased (Investigations) | 459 | 427
Neutrophil count decreased (Investigations) | 87 | 88
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 183 | 176
Cervical dysplasia (Reproductive system and breast disorders) | 94 | 118
Hypertension (Vascular disorders) | 42 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights